CLINICAL TRIAL: NCT06794060
Title: Therapeutic Effect of Vitamin C Supplementation in Patients With Ovarian Aging：a Multicenter, Double-blind, Randomized Controlled Trial
Brief Title: Therapeutic Effect of Vitamin C Supplementation in Patients With Ovarian Aging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M2024647
Record Dates: First submitted 2025-01-10; First posted 2025-01-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Premature Ovarian Insufficiency; Ovarian Reserve Function
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A double-blind design was employed for researchers were designed to be blinded. Allocation concealment was designed to apply to study subjects, clinical practitioners, outcome assessors and subsequent data analysts. The pharmaceutical company assigned numbers and labels to the drugs, and when study subjects were enrolled, they were assigned the corresponding drug number. The specific group corresponding to the number remained concealed from the project researchers, participants, and study subjects, with the blind data kept by independent personnel.
  After the follow-up, independent personnel who maintained the blind data provided group information to the data analysts. The synthetic vitamin C, natural vitamin C and control groups were still represented as A, B and C, concealing the specific identities of the ABC groups from the data analysts. After the data comparison between the two groups the unblinding of the AB groups was conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Synthetic vitamin C (Experimental): Participants will take the synthetic vitamin C twice a day, 500mg per time.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Natural vitamin C (Experimental): Participants will take the natural vitamin C twice a day, 500mg per time.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Placebo (Placebo Comparator): Participants will take tablets with the same texture, flavor, and appearance as the experimental group twice a day, 500mg per time.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C (Ascorbic Acid) — Participants swallow synthetic vitamin C tablets 500mg with water, twice a day.
  Arms: Synthetic vitamin C
Dietary Supplement: Vitamin C (Ascorbic Acid) — Participants swallow naturral vitamin C tablets 500mg with water, twice a day.
  Arms: Natural vitamin C
Other: Placebo — Participants swallow tablets with the same texture, flavor, and appearance as the experimental group 500mg with water, twice a day.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Vitamin C works to improve ovarian reserve in women with ovarian aging. It will also learn about the safety of Vitamin C. The main questions it aims to answer are:

* Does Vitamin C supplementation improve the ovarian reserve prediction score?
* What medical problems do participants have when taking Vitamin C supplementation?

Researchers will compare Vitamin C to a placebo (a look-alike substance that contains no drug) to see if drug Vitamin C works to improve ovarian reserve in women with ovarian aging. Participants will:

* Take Vitamin C or a placebo every day for 12 months
* Visit the clinic once every 4 weeks for follow-up and drug distribution.
* Return the Vitamin C box at each visit.
* Report any adverse effects of treatment to the doctor.
* Fill out a questionnaire at each visit.
* After 6 months and 12 months of intervention, take blood test and ultrasonic examination.

ELIGIBILITY:
Inclusion Criteria:

* Regularity of menstruation changed for less than one year.
* 10U/L≤ FSH<25 U/L in two tests more than 4weeks aprt.
* AMH < 1.1 ng/mL.
* Bilateral ovarian AFC <7.
* Signed informed consent and can participate in regular follow-ups.

Exclusion Criteria:

* Ovarian aging caused by TUNER (X deletion) syndrome or gene mutation.
* Ovarian aging caused by ovarian surgery or chemotherapy.
* Patients with severe endocrine system diseases (diabetes, thyroid disease), digestive system diseases (affecting VC absorption), cardiovascular system diseases, renal insufficiency (abnormal urine, imaging diagnosis, blood, pathological analysis confirms that kidney damage does exist, or glomerular filtration rate GFR <60mL/min), nervous system diseases such as dementia and epilepsy; patients with infectious diseases such as HIV, hepatitis, tuberculosis; patients with severe autoimmune diseases.
* Continuous alcohol or drug abuse (to avoid adverse reactions caused by drinking).
* Allergic to vitamin C or any component of the preparation.
* Patients who have already started large-dose (greater than 500mg/day) vitamin C supplementation.
* Unwilling to or stop taking supplements not provided by this project.
* Those who have participated in other ovarian aging clinical intervention projects.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
ovarian reserve prediction score | 1 year
  The ovarian reserve prediction score was calculated using the Ovarian Reserve Prediction Tool, OvaRePred. This tool evaluates the current ovarian reserve status and predicts the future age at which diminished ovarian reserve (DOR) and perimenopause may occur. The score ranges from 0 to 100, with higher scores indicating better ovarian function.

SECONDARY OUTCOMES:
FSH level | 1 year
  Follicle-stimulating hormone (FSH): Test the blood FSH level of women.
AMH level | 12 months
  Anti-Müllerian Hormone (AMH) is a hormone produced by the granulosa cells of ovarian follicles. It serves as a key indicator of a woman's ovarian reserve, which refers to the number of viable eggs remaining in the ovaries.
AFC | 12 months
  Antral Follicle Count (AFC), is a measure used in reproductive medicine to assess a woman's ovarian reserve, that can be seen and counted via transvaginal ultrasound.
Clinical pregnancy rate | 12 months
  A clinical pregnancy is a pregnancy that is confirmed by ultrasound.
Time to pregnancy | 12 months
  Time to pregnancy (TTP) refers to the duration it takes for a couple to conceive, starting from the time they begin trying to achieve a pregnancy.
Livebirth rate | 12 months
  A live birth refers to the delivery of a baby who shows any signs of life after being born, regardless of the pregnancy's duration.

IPD SHARING:
Plan to Share IPD: No
We have decided not to share the IPD from this study due to concerns about participant privacy and confidentiality. Despite efforts to de-identify the data, there remains a risk of re-identification, which could compromise the privacy of the participants involved. Additionally, there are legal and ethical considerations that restrict the sharing of sensitive health information without explicit consent from the participants. Furthermore, the resources required to prepare and manage the data for external sharing are currently beyond our capacity. Therefore, to ensure the protection of our participants and comply with ethical standards, we have opted not to share the IPD at this time.